CLINICAL TRIAL: NCT06231095
Title: Does TMS Affect Neuroplasticity? The Role of Brain-derived Neurotrophic Factor and Neuronal Cell Adhesion Molecules - an Intensive Clinical Protocol Among Patients With Obsessive-compulsive Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Julian Maciaszek, Principal Investigator, Wroclaw Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUBK.C230.23.065
Record Dates: First submitted 2024-01-07; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: OCD
Keywords: TMS; OCD; cTBS; BDNF; Neuroplasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: continuous theta burst stimulation - cTBS — Continuous theta burst stimulation (cTBS) is a quicker and potentially more effective technique to reduce cortical hyperactivity than repetitive transcranial magnetic stimulation (rTMS). The study involves a cycle of 35 cTBS stimulations in the supplementary motor area (SMA) over 5 working days, with 7 stimulation sessions each day lasting 40 seconds. A 1-hour break between sessions will be observed, and each session will comprise 600 pulses at 90% of the motor threshold intensity.

SUMMARY:
Patients expressing interest in participating will undergo psychiatric assessment to verify the diagnosis of treatment-resistant obsessive-compulsive disorder (OCD), assess symptom severity, and exclude TMS contraindications. The study involves a cycle of 35 continuous theta burst stimulations (cTBS) in the supplementary motor area (SMA) over 5 working days, with 7 stimulation sessions each day lasting 40 seconds. A 1-hour break between sessions will be observed, and each session will comprise 600 pulses at 90% of the motor threshold intensity.

Biochemical analysis of blood serum from 40 patients will be conducted at three time points in an open-label study with active TMS stimulation:

T0 - before starting stimulation T1 - after completing stimulation T2 - 1 month after completing stimulation

Inclusion criteria: Diagnosis of depression or OCD according to the 10th revision of the International Statistical Classification of Diseases and Related Health Problems (ICD-10) criteria, Hamilton Depression Rating Scale (HAM-D) score > 16 points, or Yale-Brown Obsessive Compulsive Scale (Y-BOCS) score > 19 points; age 18-70 years.

Exclusion criteria: Contraindications to TMS procedures, lack of informed consent, and documented persistent non-cooperation with treatment

DETAILED DESCRIPTION:
Transcranial Magnetic Stimulation (TMS) is an accepted non-invasive method of neurostimulation. Evidence has demonstrated that TMS allows for the reduction of depression symptoms, and an increasing number of reports support its efficacy in reducing symptoms of obsessive-compulsive disorder (OCD). There is a limited body of clinical research available on the mechanisms of TMS action. Neuroplasticity refers to the capacity of neural tissue to form new connections for the purpose of reorganization and adaptation. Brain-Derived Neurotrophic Factor (BDNF) and Cell Adhesion Molecules (CAM) are markers of neuroplasticity. BDNF influences transmission in both excitatory and inhibitory synapses, enhancing neurotransmitter release in cholinergic and dopaminergic neurons. According to the neurotrophic hypothesis, stress may decrease BDNF levels. Serum BDNF concentrations are reduced in untreated patients with depression and normalized by antidepressant treatment. Neuronal CAMs are among the most prevalent proteins, playing a crucial role in synaptic plasticity. Various CAMs appear to interact with BDNF. In depression, both reduced BDNF levels and polysialylated (PSA) neuronal CAMs are observed. Conversely, the levels of Vascular Cell Adhesion Molecule-1 (VCAM-1) and Intracellular Adhesion Molecule-1 (ICAM-1) in depression are inversely correlated with BDNF.

To address this gap, the investiagators aimed to verify the hypothesis that TMS in OCD leads to symptom reduction by inducing neuroplasticity through:

Comparing changes in BDNF and CAM protein concentrations after TMS stimulation in OCD patients before and after stimulation.

Assessing the correlation between changes in BDNF and CAM concentrations and the reduction of psychopathological symptoms.

Evaluating the predictive value of initial BDNF and CAM concentrations.

Study assumptions and planned procedures:

Patients expressing interest in participating will undergo psychiatric assessment to verify the diagnosis of treatment-resistant OCD, assess symptom severity, and exclude TMS contraindications. The study involves a cycle of 35 cTBS stimulations in the supplementary motor area (SMA) over 5 working days, with 7 TMS sessions each day lasting 40 seconds. A 1-hour break between sessions will be observed, and each session will comprise 600 pulses at 90% of the motor threshold intensity.

Biochemical analysis of blood serum from 40 patients will be conducted at three time points in an open-label study with active TMS stimulation:

T0 - before starting stimulation T1 - after completing stimulation T2 - 1 month after completing stimulation

Inclusion criteria: Diagnosis of depression or OCD according to ICD-10 criteria, Hamilton Depression Rating Scale (HAM-D) score > 16 points, or Yale-Brown Obsessive Compulsive Scale (Y-BOCS) score > 19 points; age 18-70 years.

Exclusion criteria: Contraindications to TMS procedures, lack of informed consent, and documented persistent non-cooperation with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of depression or OCD according to ICD-10 criteria,
* Yale-Brown Obsessive Compulsive Scale (Y-BOCS) score > 19 points;
* age 18-70 years.

Exclusion Criteria:

* Contraindications to TMS procedures,
* lack of informed consent, and documented persistent non-cooperation with treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2024-01-06 (Actual)

PRIMARY OUTCOMES:
OCD symptoms severity T1 | 5 days
  OCD symptoms severity - Yale Brown Obsessive-Compulsive Scale (Y-BOCS) scoring from 0-40. Higher score means higher severity of symptoms
OCD symptoms severity T2 | 30 days
  OCD symptoms severity - OCD symptoms severity - Yale Brown Obsessive-Compulsive Scale (Y-BOCS) scoring from 0-40. Higher score means higher severity of symptoms
depressive symptoms severity T1 | 5 days
  depressive symptoms severity -Montgomery-Asberg Depression Rating Scale (MADRS) scoring from 0-60. Higher score means higher severity of depressive symptoms
depressive symptoms severity T2 | 30days
  depressive symptoms severity - depressive symptoms severity -Montgomery-Asberg Depression Rating Scale (MADRS) scoring from 0-60. Higher score means higher severity of depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Błażej Misiak, Prof, Study Chair — Department of Psychaitry Wroclaw Medical Univeristy, Pasteura 10 Str Wrocław Poland
Locations (2):
- Poland (2):
  - Department of Psychaitry Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship
  - Deprtment of Psychiatry, Wroclaw, Lower Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: No